CLINICAL TRIAL: NCT05733767
Title: Implementing Effective Smoking Cessation Pharmacotherapy for Hospitalized Smokers With Cardiopulmonary Disease
Brief Title: Smoking Cessation Pharmacotherapy-Nurse Practitioner Led Tobacco Treatment Team Study
Acronym: STOP-NPT3
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Collaborators: University of Massachusetts Chan Medical School, Worcester (Unknown); Boston University (Other); University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL15685
Record Dates: First submitted 2023-01-05; First posted 2023-02-17 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-02

CONDITIONS: Cardiopulmonary Disease; Smoking Cessation; Inpatient
MeSH Terms: conditions — Pulmonary Heart Disease; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced usual care (EUC) (Active Comparator): The investigators will administer the enhanced usual care intervention to randomized patients.
  Interventions: Other: Enhanced Usual Care (EUC)
- Personalized Care: Nurse Practitioner led Tobacco Treatment Team (NPT3) (Experimental): The investigators will administer the personalized care NPT3 intervention to randomized patients.
  Interventions: Other: Nurse Practitioner Tobacco Treatment Team (NPT3)

INTERVENTIONS:
Other: Enhanced Usual Care (EUC) — Patients randomized to arm 1, enhanced care (EC), will receive the following intervention: 1) referral to the state quitline, 1-800-QUIT-NOW, 2) primary care physician notification of an ongoing quit attempt, and 3) enrolled in an assessment-only text message system. This text message system will assess medication use and self-reported smoking cessation outcomes, but will not provide any counseling, advice, or feedback. Participants in arm 1 will receive a text message at discharge, and then they will receive 1 text assessment at the following time points: day 7, month 1, and month 3.
  Arms: Enhanced usual care (EUC)
Other: Nurse Practitioner Tobacco Treatment Team (NPT3) — Patients randomized to arm 2, personalized care (PC), will receive a multi-component, multi-disciplinary smoking cessation intervention in addition to usual care. This intervention will include three main interventions. First, a nurse practitioner will assess all patients and then prescribe tailored medications for smoking cessation based on patient preferences. Patients will also then receive a sample ad-lib nicotine replacement therapy (NRT) packet for use as needed to their prescribed medications. Second, a Tobacco Treatment Counselor (TTC) will provide personalized advice, education, and coaching to the patient and encourage medication adherence. Third, patients will be enrolled in a smoking cessation text messaging program designed to maintain motivation, encourage medication adherence, and allow communication with the team. The text message program will last for 6 months and will include assessment at the following time points: day 7, month 1, and month 3.
  Arms: Personalized Care: Nurse Practitioner led Tobacco Treatment Team (NPT3)

SUMMARY:
Tobacco use remains the leading cause of death in the United States and contributes to more than 7 million hospitalizations annually. Being admitted to the hospital offers the perfect opportunity to support smoking cessation. Patients are motivated to quit because of their current illness and societal guidelines recommend clinicians should counsel patients and prescribe smoking cessation pharmacotherapy (SCP) to virtually all smokers.

However, only 22% of patients are prescribed SCP while hospitalized, and only 1% are prescribed medications compatible with current guidelines. This failure is part of the reason 70-80% of hospitalized smokers eventually relapse. The relapse typically occurs within a few days of hospital discharge - well before outpatient follow-up can occur.

The investigators aim to improve smoking cessation treatment and guideline adherence by utilizing the opportunity that hospitalization provides. The investigators have created a tobacco treatment team (T3) to overcome physicians' and patients' low use of current guideline smoking cessation medications. The team members are trained in tobacco treatment and will be led by a nurse practitioner (NPT3). The team will work together and 1) prescribe individually tailored and guideline-concordant SCP; 2) counsel and motivate patients to use SCP properly; and 3) manage a mobile phone-based text-messaging system to keep patients motivated and adherent to SCP. Our preliminary data suggest that such an approach is workable and acceptable to patients, physicians, and hospital administrators.

The investigators will recruit 424 patients in the hospital who smoke with cardiopulmonary disease. These patients will be randomized to receive either usual care or personalized care with the NPT3 team. The investigators will compare rates of guideline-concordant SCP use at 1 week and exhaled carbon monoxide (eCO) verified smoking cessation at 6 months between patients randomized to the NPT3 team vs. usual care.

The investigators will also measure the project's economic value from a hospital and payer perspective. Understanding the economic value will better inform hospital and insurance policies and sustainability. Finally, acceptability, generalizability, and sustainability measures will be assessed through qualitative interviews with patients, providers, and hospital leadership.

DETAILED DESCRIPTION:
This study aims to conduct a single-center, type 2, hybrid implementation-effectiveness trial, evaluating a strategy for improving prescription and uptake of smoking cessation pharmacotherapy (SCP) among smokers hospitalized for a cardiopulmonary condition. Patients will be recruited at Baystate Medical Center, Springfield MA from an electronic medical record (EMR) alert upon hospital admission indicating the patient smokes cigarettes. The investigators will then screen the EMR, and those who pass the EMR screen will be introduced to the study. Eligible, consenting patients will be randomized to one of two study arms: 1) Enhanced Usual Care (EUC) or 2) Nurse Practitioner led-Tobacco Treatment Team (NPT3) intervention. Randomization will be stratified by current smoking status (< 10 / 10+ cigarettes/day).

The investigators will evaluate the following primary implementation hypothesis: Patients randomized to the NPT3 intervention will be more likely to use guideline-concordant smoking cessation medications 7 days after hospital discharge compared to patients randomized to EUC. The primary effectiveness hypothesis is: Patients randomized to the intervention group will be more likely to quit smoking at 6 months. The investigators will evaluate the use of guideline-concordant SCP as a mediator of quit status at 6 months.

The investigators will recruit 424 patients to participate in the main clinical trial of enhanced usual care compared to the multi-component tobacco treatment team, NPT3 (Aim 1). These patients will be assessed at baseline and followed for 6 months for outcomes. Clinical outcomes will be collected up to 3 years after trial participation.

The investigators, proposed sample (n= 424 total patients) has 90% power to detect a clinically meaningful 15% improvement in smoking cessation rates at 6 months and a 99% power to detect a significant difference in guideline-concordant medication use at 1 week post-hospital discharge. A 20% smaller sample (n=340), due to low recruitment or attrition, would still achieve >80% power to find the intervention different from the control.

All analyses will be performed using an intent-to-treat approach, based upon the randomization arm, regardless of adherence to the intervention. The investigators will use logistic regression models to estimate the effect of the study arm (NPT3 vs. EUC), which will include randomization stratum and unbalanced baseline characteristics (if any.) In addition, the investigators will explore sex and socioeconomic status (SES) as modifiers of guideline-concordant SCP use and smoking cessation outcomes by including sex-by-study-arm and SES-by-study arm interaction terms. Missing data will be analyzed for patterns of missingness and imputed in sensitivity analyses as appropriate. Finally, the investigators will perform a mediation analysis to estimate the independent impact of SCP on smoking cessation outcomes.

The investigators will monitor for adverse events. All adverse events/effects will be recorded in the research record, and any reports of adverse events will be reviewed by the PI or their designees, who are available 24 hours a day. All non-serious adverse events will be reviewed in a weekly study meeting. Adverse event documentation will include a description of the event, ratings of severity and relationship to study procedures, follow-up (if any), and outcome. All serious and non-serious adverse events will be summarized in the required report to the institutional review board (IRB) and data safety monitoring board (DSMB).

ELIGIBILITY:
Inclusion Criteria:

* Admitted to Baystate Medical Center in Springfield, MA with a cardiac or pulmonary disease diagnosis will be eligible to participate in this trial.
* Patients who smoke cigarettes
* Speak English

We will include any patients with the following diagnoses or procedures from Baystate Medical Center in Springfield, MA:

* myocardial infarction
* coronary artery bypass grafting surgery
* heart valve surgery
* percutaneous coronary intervention (PCI)
* acute coronary syndrome
* heart failure
* chronic obstructive pulmonary disease (COPD)
* asthma exacerbation.

Exclusion Criteria:

* We will exclude pregnant or nursing women, patients with current suicidal ideation, planned discharge to hospice or expected survival <6 months, or concurrent use of daily smoked marijuana, because this can increase exhaled carbon monoxide levels, which would confound biochemical confirmation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2027-08-28 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients using guideline concordant smoking cessation medication at 7 days | 7 days after hospital discharge
  Use of varenicline or combination medications (nicotine patch and lozenge, gum, or inhaler) on the 7th day after discharge
Proportion of patients reporting smoking cessation abstinence (7 day point prevalence at 6 months) | 7 day point prevalence at 6 months after hospital discharge
  Patients who have self-reported not using any tobacco products in the 7 days prior to assessment, then confirmed with an in-office exhaled carbon monoxide level of <6 ppm.

SECONDARY OUTCOMES:
Proportion of patients using guideline concordant smoking cessation medication throughout the study time frame. | Day -1 (at consent and while admitted), Day 0 (Discharge day), Day 30 (1 month after discharge), Day 90 (3 months after discharge), Day 180 (6 months after discharge)
  Use of varenicline or combination of medications (bupropion, nicotine patch, lozenge, gum, or inhaler) at these time points
Proportion of patients using any smoking cessation medication throughout study time frame | Day -1 (at consent and while admitted), Day 0 (Discharge day), Day 30 (1 month after discharge), Day 90 (3 months after discharge), Day 180 (6 months after discharge)
  Use of any smoking cessation medication (bupropion, nicotine patch, lozenge, gum, or inhaler) at these time points
Proportion of patients reporting smoking cessation abstinence (7 day point prevalence at 7 days, 30days, and 90 days post- discharge) | 7 day point-prevalence: a. 7 days after hospital discharge b. 1 month after discharge c. 3 months after discharge
  Patients who have self-reported not using any tobacco products in the 7 days prior to assessment at these time points
Proportion of patients reporting continuous abstinence smoking cessation | Continuous abstinence: a. 1 month after discharge b. 3 months after discharge c. 6 months after discharge
  Patients who have self-reported not using any tobacco products since hospital discharge

OTHER OUTCOMES:
Proportion of patients reporting a hospital readmission throughout the study time frame | Within 30 days, 3 months, and 6 months after hospital discharge
  Patients who are admitted to the hospital (full admission or observation status) with apparent life-threatening illness
Proportion of patients reporting medication side effects and cumulative medication side effects reported | Within 6 months after hospital discharge
  Any reported side-effects to medications including but not limited to nausea, abnormal dreams, rash, insomnia, dyspepsia, hiccups, headache, and seizures.
Proportion of patients reporting E-cigarette use | At 6 months after hospital discharge
  Patients who endorse using any form of e- cigarettes
Proportion of patients reporting number of quit attempts | Within 6 months after hospital discharge
  Quit attempt is defined as going >24 hours without a cigarette in an attempt to quit; this includes the hospital-based baseline quit attempt
Longest period of continuous abstinence | Within 6 months after hospital discharge
  The longest period of self-reported abstinence without a single cigarette, as measured in weeks
Cigarettes smoked per day | At 6 months after hospital discharge
  The number of self-reported cigarettes smoked per day

CONTACTS AND LOCATIONS:
Overall Officials: Quinn R Pack, MD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No